CLINICAL TRIAL: NCT04035577
Title: Expanding College Student Mental Health With Stress Management Mobile Technologies - Extended Usability Trial
Brief Title: IntelliCare in College Students
Acronym: ICCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Emily G Lattie, Assistant Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: K08MH112878-EUT; K08MH112878 (NIH)
Record Dates: First submitted 2019-07-23; First posted 2019-07-29 (Actual); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Depression; Anxiety
Keywords: Mental health; App; Mobile phone; Stress management
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Mobile self-help intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Extended usability of a mobile self-help intervention (Experimental): Participants will have open access to the Intellicare Hub app for 8-weeks and be surveyed at Baseline, 4-weeks, and 8-weeks
  Interventions: Behavioral: Mobile self-help intervention

INTERVENTIONS:
Behavioral: Mobile self-help intervention — During the trial, participants will use Intellicare apps for up to 8 weeks and will be invited to provide feedback about their experience at two follow-up time points: weeks 4 and 8. All participants will first undergo initial assessments that will include a series of online questionnaires about their mood. Eligible participants will receive up to 8 weeks of access to the IntelliCare system, which consists of apps with a variety of resources, including lessons and tools designed to teach skills for mood management. It is suggested that participants utilize the mobile phone tools every day

SUMMARY:
This study is an 8-week usability and feasibility trial of the smartphone student stress-management app IntelliCare for college students. This intervention will be tested with University of Illinois at Chicago (UIC) and Northern Illinois University (NIU) students. During this period, research surveys assessing depression and anxiety can be completed on the app. Also, user feedback interviews will be conducted viatelephone at four weeks and at eight weeks to gain insight on the user experience of IntelliCare for College Students.

DETAILED DESCRIPTION:
In this study, students will be recruited for an 8-week trial in which they will be given the IntelliCare Hub app and encouraged to use it daily. To ensure a sample representative of likely end users, 10 students from each site will be recruited: 5 with elevated distress as measured by scores > 10 on either the PHQ-9 or GAD-7 and 5 without elevated scores on either measure, for a total of 20 participants. The rationale for 10 participants in each group is based on past usability research indicating saturation is typically reached within 10 participants. This trial aims to identify software bugs and usability problems that emerge over extended use and to examine preliminary effects of program use. During the trial, participants will be prompted to complete the PHQ-8 and GAD-7 every week. At baseline, 4 weeks, and 8 weeks, participants will be prompted within the app to complete the Depression Literacy Questionnaire and Anxiety Literacy Questionnaire to measure mental health literacy, the Knowledge and Beliefs about Services scale to measure knowledge of campus mental health services, the Barriers to Mental Health Help-Seeking questionnaire to measure treatment barriers, and the Cognitive and Behavioral Response to Stress Scale to measure cognitive and behavioral coping skills. At 4 and 8 weeks participants will be asked to participate in a user-feedback interview via the telephone. This is to gain insight on the user's experience with the app.

ELIGIBILITY:
Inclusion Criteria:

Participant is a student at the University of Illinois in Chicago or Northern Illinois University. Participant owns a smartphone capable of running Android 7 (or higher) or iOS11 (or higher).

Participant is 18 years of age or older

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lattie E, Cohen KA, Winquist N, Mohr DC. Examining an App-Based Mental Health Self-Care Program, IntelliCare for College Students: Single-Arm Pilot Study. JMIR Ment Health. 2020 Oct 10;7(10):e21075. doi: 10.2196/21075. PMID 33037874

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant withdrew from the study after signing the consent form but before initiating any of the study activities, and we consented an additional participant in their place. A total of 21 participants consented.
Period: Overall Study
Arm/Group | Extended Usability of a Mobile Self-help Intervention
Started | 21 (One participant withdrew after signing the consent but before initiating any study activities.)
Completed | 19
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Extended Usability of a Mobile Self-help Intervention
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.19 (6.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 7
  More than one race | 6
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 21
Patient Health Questionnaire - 8 (PHQ-8) - Depression Severity Module [Mean (Standard Deviation); unit: units on a scale] — The PHQ-8 measures degree of depression severity. Possible range of scores for the PHQ-8 is 0-24. Higher values represent a worse outcome.
  Specifically, scores of 0-4 indicate minimal or no depression; 5-9 is mild; 10-14 is moderate; 15-19 is moderately severe; and 20-24 is severe.
  For the subgroups presented, participants with a score less than 10 were in the "lower symptom" subgroup, and participants with a score greater than or equal to 10 were in the "higher symptom subgroup" Population: Subgroup means are provided
  units on a scale
    Lower symptom: number analyzed (Participants) | 9
    Lower symptom | 3.75 (2.38)
    Higher symptom: number analyzed (Participants) | 11
    Higher symptom | 11.63 (6)
GAD-7 (Generalized Anxiety Disorder Scale-7) [Mean (Standard Deviation); unit: units on a scale] — The GAD-7 is a self-administered 7 item instrument that uses DSM-V criteria for GAD (General Anxiety Disorder) to measure symptom severity. GAD-7 total score for the seven items ranges from 0 to 21. Higher values represent a worse outcome. Specifically, scores of 1-4 indicate minimal anxiety symptoms; 5-9 is mild anxiety symptoms; 10-14 is moderate anxiety symptoms; and 15-21 is severe anxiety symptoms.
  Participants with a score < 10 are in the "lower symptom" subgroup. Participants with a score greater than or equal to 10 are in the "higher symptom" subgroup. Population: Subgroup means presented
  units on a scale
    Lower symptom: number analyzed (Participants) | 9
    Lower symptom | 4.88 (2.85)
    Higher symptom: number analyzed (Participants) | 11
    Higher symptom | 10.82 (4.12)
Anxiety Literacy Questionnaire [Mean (Standard Deviation); unit: units on a scale] — This questionnaire is designed to assess anxiety specific mental health literacy by presenting 22 true or false statements regarding anxiety (e.g., "Being easily fatigued may be a symptom of anxiety disorder.") Participants receive a score of 1 for each statement they correctly assign as either true or false. Scores for each questionnaire can range from 0-22, with higher scores indicating greater anxiety specific mental health literacy.
  units on a scale | 13.88 (3.67)
Depression Literacy Questionnaire [Mean (Standard Deviation); unit: units on a scale] — This questionnaire is designed to assess depression specific mental health literacy by presenting 22 true or false statements regarding anxiety and depression (e.g., "Loss of confidence and poor self-esteem may be a symptom of depression.") Participants receive a score of 1 for each statement they correctly assign as either true or false. Scores for each questionnaire can range from 0-22, with higher scores indicating greater depression specific mental health literacy
  units on a scale | 13.89 (4.29)
Cognitive and Behavioral Response to Stress Scale [Mean (Standard Deviation); unit: units on a scale] — This is an 18-item scale designed to measure the use and helpfulness of cognitive and behavioral skills. There are four subscales: cognitive skill frequency, cognitive skill usefulness, behavioral skill frequency, and behavioral skill usefulness. For each skill, participants rate how often they used it and how helpful it was. Cognitive subscales scores range from 0-24, and scores from behavioral subscales can range from 0-30. Higher scores indicate better outcomes.
  units on a scale
    CB-RSS cognitive usefulness | 9.73 (6.23)
    CB-RSS cognitive frequency | 10.47 (4.03)
    CB-RSS behavioral usefulness | 17.74 (6.10)
    CB-RSS behavioral frequency | 14.42 (4.98)

OUTCOME MEASURES:

1. Primary Outcome: Patient Health Questionnaire - 8 (PHQ-8) - Depression Severity Module
Description: The PHQ-8 measures degree of depression severity. Possible range of scores for the PHQ-8 is 0-24. Higher values represent a worse outcome.
  Specifically, scores of 0-4 indicate minimal or no depression; 5-9 is mild; 10-14 is moderate; 15-19 is moderately severe; and 20-24 is severe.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Lower Symptom: Participants who had PHQ-9 and GAD-7 scores under 10 at baseline
- Higher Symptom: Participants who had a score of 10 or greater on the PHQ-9 of GAD-7 at baseline
Arm/Group | Lower Symptom | Higher Symptom
Number analyzed (Participants) | 9 | 10
score on a scale | 2.43 (2.51) | 9.28 (2.49)

2. Primary Outcome: Patient Health Questionnaire - 8 (PHQ-8) - Depression Severity Module
Description: The PHQ-8 measures degree of depression severity. Possible range of scores for the PHQ-9 is 0-24. Higher values represent a worse outcome.
  Specifically, scores of 0-4 indicate minimal or no depression; 5-9 is mild; 10-14 is moderate; 15-19 is moderately severe; and 20-24 is severe.
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lower Symptom | Higher Symptom
Number analyzed (Participants) | 9 | 10
score on a scale | 0.6 (2.51) | 9 (6.53)

3. Primary Outcome: GAD-7 (Generalized Anxiety Disorder Scale-7)
Description: The GAD-7 is a self-administered 7 item instrument that uses some of the DSM-V criteria for GAD (General Anxiety Disorder) to identify probable cases of GAD along with measuring anxiety symptom severity. GAD-7 total score for the seven items ranges from 0 to 21. Higher values represent a worse outcome. Specifically, scores of 1-4 indicate minimal anxiety symptoms; 5-9 is mild anxiety symptoms; 10-14 is moderate anxiety symptoms; and 15-21 is severe anxiety symptoms.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lower Symptom | Higher Symptom
Number analyzed (Participants) | 9 | 10
score on a scale | 2.86 (2.61) | 10.14 (2.79)

4. Primary Outcome: GAD-7 (Generalized Anxiety Disorder Scale-7)
Description: as for outcome 3
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lower Symptom | Higher Symptom
Number analyzed (Participants) | 9 | 10
score on a scale | 2.86 (2.61) | 10 (3.83)

5. Primary Outcome: Anxiety Literacy Questionnaire
Description: This questionnaire is designed to assess anxiety specific mental health literacy by presenting 22 true or false statements regarding anxiety (e.g., "Being easily fatigued may be a symptom of anxiety disorder.") Participants receive a score of 1 for each statement they correctly assign as either true or false. Scores for each questionnaire can range from 0-22, with higher scores indicating greater anxiety specific mental health literacy.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended Usability of a Mobile Self-help Intervention
Number analyzed (Participants) | 19
score on a scale | 14 (3.32)

6. Primary Outcome: Anxiety Literacy Questionnaire
Description: as for outcome 5
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended Usability of a Mobile Self-help Intervention
Number analyzed (Participants) | 19
score on a scale | 14.63 (3.45)

7. Primary Outcome: Depression Literacy Questionnaire
Description: This questionnaire is designed to assess depression specific mental health literacy by presenting 22 true or false statements regarding anxiety and depression (e.g., "Loss of confidence and poor self-esteem may be a symptom of depression.") Participants receive a score of 1 for each statement they correctly assign as either true or false. Scores for each questionnaire can range from 0-22, with higher scores indicating greater depression specific mental health literacy
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended Usability of a Mobile Self-help Intervention
Number analyzed (Participants) | 19
score on a scale | 14.5 (3.97)

8. Primary Outcome: Depression Literacy Questionnaire
Description: as for outcome 7
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended Usability of a Mobile Self-help Intervention
Number analyzed (Participants) | 19
score on a scale | 14.68 (3.83)

9. Primary Outcome: Cognitive and Behavioral Response to Stress Scale
Description: This is an 18-item scale designed to measure the use and helpfulness of various cognitive and behavioral skills. There are four subscales included: cognitive skill frequency, cognitive skill usefulness, behavioral skill frequency, and behavioral skill usefulness. For each cognitive or behavioral skill, participants rate how often they used the skill and how helpful it was (e.g. "During the past month, how often did you take a moment to notice things that made you feel good or grateful? How helpful was this in making you feel better?"). Scores for cognitive subscales range from 0-24, and scores from behavioral subscales can range from 0-30. Higher scores indicate better outcomes.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended Usability of a Mobile Self-help Intervention
Number analyzed (Participants) | 19
score on a scale
  CB-RSS cognitive usefulness | 12.22 (6.53)
  CB-RSS cognitive frequency | 11.55 (5.03)
  CB-RSS behavioral usefulness | 19.22 (7.38)
  CB-RSS behavioral frequency | 15.72 (7.20)

10. Primary Outcome: The Cognitive and Behavioral Response to Stress Scale
Description: as for outcome 9
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended Usability of a Mobile Self-help Intervention
Number analyzed (Participants) | 19
score on a scale
  CB-RSS cognitive usefulness | 12.58 (6.86)
  CB-RSS cognitive frequency | 12.68 (4.49)
  CB-RSS behavioral usefulness | 19.68 (8.91)
  CB-RSS behavioral frequency | 16.52 (6.44)

11. Secondary Outcome: Mean Number of Treatment App Use Sessions
Time Frame: Daily for two months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Extended Usability of a Mobile Self-help Intervention
Number analyzed (Participants) | 19
days | 17.05 (8.12)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Extended Usability of a Mobile Self-help Intervention
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2019-06-16): https://cdn.clinicaltrials.gov/large-docs/77/NCT04035577/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/77/NCT04035577/Prot_SAP_001.pdf